CLINICAL TRIAL: NCT05051046
Title: Colorectal Cancer Screnning Colonoscopy Under Hypnosis: A Multicenter Randomized Non-Inferiority Trial
Brief Title: Colorectal Cancer Screnning Colonoscopy Under Hypnosis
Acronym: CODEPICCH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: DR200072
Record Dates: First submitted 2021-07-20; First posted 2021-09-21 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Colorectal (Colon or Rectal) Cancer
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypnosis (Experimental)
  Interventions: Procedure: Colonoscopy under hypnosis
- General anesthesia (No Intervention): Common practice

INTERVENTIONS:
Procedure: Colonoscopy under hypnosis — The hypnosis used will be of the Ericksonian type. Before the colonoscopy begins, the IDE puts the patient in a hypnotic situation.
  Arms: Hypnosis

SUMMARY:
Through this study, the effectiveness of hypnosis in the realization of a colonoscopy for the detection of colorectal cancer will be evaluated

DETAILED DESCRIPTION:
Colorectal cancer is the 3rd most common cancer. Colonoscopy, a screening examination, has led to an increase in patient survival. In more than 90% of cases, this examination is performed under general anesthesia (GA) because it is considered painful, even though several studies have shown its feasibility without GA with a good tolerance in 75% of cases. However, only 28% of patients accept the examination without GA because of great apprehension. GA entails an increased risk of complications but also additional costs. Thus, performing colonoscopies without GA would reduce risks and costs by 15 to 30%. In order to make the examination more acceptable and less anxiety-provoking, methods such as hypnosis have been tested with the result that pain and anxiety are reduced and the hemodynamic state of the patients is stabilized, thus reducing the examination time. To date, the majority of studies on hypnosis, of varying indications, are small, mono-centric and non-randomized.

The use of hypnosis for colorectal cancer screening colonoscopies would reduce patient anxiety, avoid complications related to GA and reduce the organizational constraints and costs related to GA.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age or older
* Undergoing a screening colonoscopy (mass screening Fecal Immunochemical Test positive or as an individual (family history of colon cancer or adenoma, personal history of adenoma, cancer, chronic inflammatory bowel disease) or in the context of a transit disorder, hemorrhage or anemia
* Affiliated with a French social security system
* Having signed a written consent

Exclusion Criteria:

* Patient requiring emergency colonoscopy
* History of colonic resection
* Carriers of behavioral disorders and/or psychiatric illness
* Limited cognitive abilities making it impossible to read or fill out a discrete choice questionnaire (language problems, comprehension problems)
* Contraindication to hypnosis, preventing quality interaction (comprehension and/or language problems, hearing impairment)
* Contraindication to general anesthesia
* Under a legal protection regime
* Pregnant or breastfeeding woman

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2022-01-31 (Actual); Primary Completion 2028-02-07 (Estimated); Study Completion 2028-02-07 (Estimated)

PRIMARY OUTCOMES:
Rate of complete colonoscopies | The day of the colonoscopy, from the start to the end of the colonoscopy
  Rate of complete colonoscopies: a colonoscopy is said to be complete when the endoscopist visualizes the caecal fundus.

SECONDARY OUTCOMES:
Level of anxiety | The day of the colonoscopy, before the exam
  Level of anxiety is measured by the State-Trait Anxiety Inventory (Form Y) scale
Level of pain | During the consultation before the colonoscopy
  pain level measured by self-evaluation via a visual analog scale between 0 and 10 cm, at the consultation, before and after the colonoscopy in both groups and during the procedure, before returning to the room only in the Hypnosis group. The doctor will present the ungraded side of the VAS to the patient and ask him/her to place the cursor on the maximum pain intensity felt during the procedure.
Level of pain | Up to 24 hours the day of colonoscopy
  pain level measured by self-evaluation via a visual analog scale between 0 and 10 cm, at the consultation, before and after the colonoscopy in both groups and during the procedure, before returning to the room only in the Hypnosis group. The doctor will present the ungraded side of the VAS to the patient and ask him/her to place the cursor on the maximum pain intensity felt during the procedure.
Duration of colonoscopy | The day of colonoscopy from the start to the end of the exam
  Duration of the endoscopy measured in minutes, distinguishing between: the time between the introduction of the endoscope into the anus and its arrival at the caecal floor and the time required in the opposite direction. The time taken to remove the polyps will be counted.
Rate of polyps resected | The day of colonoscopy from the start to the end of the exam
  compare the rate of resected polyps between the two groups
Rate of complications | To the day of the exam to 8 days after
  Rate of complications within 8 days post-colonoscopy (perforation, bleeding, inhalation pneumonitis, ...). Patients will be instructed to call back the service in case of complications
Patient satisfaction | Up to 24 hours the day of the colonoscopy
  Patient satisfaction questionnaire regarding the different stages of their care as well as their future wishes regarding the procedure to be considered in the event of a new colonoscopy. The satisfaction questionnaire will focus on the patient's experience of the management on arrival, the set-up in the examination room and the procedure. The best way to verify patient satisfaction is to ask the patient if he or she would like the next colonoscopy to be done under the same conditions.
Medico economic criteria | To the day of the exam to 3 months after
  Proportion of pairs (Δ cost, Δ effect) belonging to the non-inferiority area in the incremental cost-effectiveness design, for different values of the economic non-inferiority margin and at constant value of the clinical non-inferiority margin (5%).

CONTACTS AND LOCATIONS:
Overall Officials: Driffa MOUSSATA, PhD, Principal Investigator — University Hospital Center of Tours
Locations (1):
- Chu Angers, Angers, France

IPD SHARING:
Plan to Share IPD: No